CLINICAL TRIAL: NCT00001001
Title: A Clinical Study Examining the Pharmacokinetics and Bioavailability of Azidothymidine (AZT, Zidovudine) in Patients With Human Immunodeficiency Virus (HIV) Infection and Hepatic Disease
Brief Title: A Study of Zidovudine in HIV-Infected Patients With Liver Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: ACTG 062; 11036 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Liver Diseases
Keywords: Liver; Liver Diseases; Liver Function Tests; HIV Seropositivity; Acquired Immunodeficiency Syndrome; Zidovudine; Biological Availability
MeSH Terms: conditions — HIV Infections; Liver Diseases; HIV Seropositivity; Acquired Immunodeficiency Syndrome | interventions — Zidovudine

INTERVENTIONS:
Drug: Zidovudine

SUMMARY:
To examine the pharmacokinetics (blood levels) and bioavailability of zidovudine (AZT) given to patients with HIV infection and chronic liver disease. The specific aim of the study is to provide data permitting the development of guidelines for use of AZT in patients with mild, moderate, or severe liver disease.

AZT is the only antiviral agent that has been shown to be effective in patients with severe HIV infection. However, AZT is largely eliminated from the body through a biochemical reaction that takes place in the liver, and it is possible that patients with underlying liver disease may have altered AZT pharmacokinetics and may metabolize AZT differently, with the result that they are susceptible to an increased risk of serious drug toxicity. This study will examine the pharmacokinetics, elimination, and metabolism of AZT in patients with liver disease. Guidelines developed from the data will be helpful in managing AZT treatment of these HIV-infected persons and will indicate whether the dose of AZT administered should be adjusted to compensate for any changes in its bioavailability and/or pharmacokinetics.

DETAILED DESCRIPTION:
AZT is the only antiviral agent that has been shown to be effective in patients with severe HIV infection. However, AZT is largely eliminated from the body through a biochemical reaction that takes place in the liver, and it is possible that patients with underlying liver disease may have altered AZT pharmacokinetics and may metabolize AZT differently, with the result that they are susceptible to an increased risk of serious drug toxicity. This study will examine the pharmacokinetics, elimination, and metabolism of AZT in patients with liver disease. Guidelines developed from the data will be helpful in managing AZT treatment of these HIV-infected persons and will indicate whether the dose of AZT administered should be adjusted to compensate for any changes in its bioavailability and/or pharmacokinetics.

Patients are assessed and stratified according to liver function and severity of liver disease. Patients receive an intravenous (IV) dose of AZT on the first day of the study, followed by an oral dose 24 hours later on the second day of the study. Patients fast for 8 hours prior to each dose and for 2 hours after each dose. Liver function tests are repeated on the first day of the study. In each patient, serial measurements of serum and urine AZT and its metabolite, 3'-azido-3'-deoxy-5'-glucuronylthymidine (GAZT), are monitored after both doses.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed after completion of day 2 of study:

* Prior medications may be resumed.

Concurrent Treatment:

Allowed after completion of day 2 of study:

* Cytotoxic chemotherapy or radiation therapy for Kaposi's sarcoma.

The study will be divided into three groups of cooperative patients according to mild, moderate, or severe liver disease. Severity of disease will be assessed within 7 days of entry into the study according to laboratory values. Patients must have normal kidney function. No medications should be taken for 48 hours prior to entering the study. Hemophiliacs are included.

Prior Medication:

Allowed:

* Zidovudine (AZT) if discontinued at least 48 hours prior to study entry.

Exclusion Criteria

Co-existing Condition:

Patients will be excluded from the study if unacceptable toxicity develops or if an illness requiring concurrent treatment develops.

Concurrent Medication:

Excluded within 48 hours of study entry:

* All medications. Medication may be resumed after completion of day 2 of the study.

Concurrent Treatment:

Excluded within 48 hours of study entry:

* All treatments. Treatment may be resumed after completion of day 2 of the study.

Patients will be excluded for the following reasons:

* Presence of active opportunistic infections, with the exception of active or chronic hepatitis B virus or hepatitis D virus infection, or ongoing therapy for an opportunistic infection.
* Thrombocytopenia, with platelets less than 50000 platelets/mm3.
* Neutropenia, with polymorphonuclear leukocytes less than 1000 cells/mm3.
* Renal insufficiency, with creatinine greater than 1.5 mg/dl.
* Acute viral hepatitis within 30 days of the study.
* Patients who are expected to be noncompliant or who are unwilling to sign an informed consent statement.

Prior Medication:

Excluded within 48 hours of study entry:

* All medications. Medication may be resumed after completion of day 2 of the study.

Prior Treatment:

Excluded within 30 days of study entry:

* Cytotoxic chemotherapy or radiation therapy for Kaposi's sarcoma. Treatment may be resumed after completion of day 2 of the study.

Active drug or alcohol abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39
Dates: Study Completion 1990-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lemon SM, Study Chair
Locations (5):
- United States (5):
  - Boston Med Ctr, Boston, Massachusetts
  - Univ of Massachusetts Med Ctr, Worcester, Massachusetts
  - Univ of North Carolina, Chapel Hill, North Carolina
  - Milton S Hershey Med Ctr, Hershey, Pennsylvania
  - Univ of Washington, Seattle, Washington

REFERENCES:
- [Background] Moore KH, Raasch RH, Brouwer KL, Opheim K, Cheeseman SH, Eyster E, Lemon SM, van der Horst CM. Pharmacokinetics and bioavailability of zidovudine and its glucuronidated metabolite in patients with human immunodeficiency virus infection and hepatic disease (AIDS Clinical Trials Group protocol 062). Antimicrob Agents Chemother. 1995 Dec;39(12):2732-7. doi: 10.1128/AAC.39.12.2732. PMID 8593010